CLINICAL TRIAL: NCT00912587
Title: Effect of Ghrelin on Sympathetic Nervous System and Stress Reactivity
Brief Title: Effect of Ghrelin on Sympathetic Nervous System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baker Heart and Diabetes Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2009/119; 11/09
Record Dates: First submitted 2009-06-01; First posted 2009-06-03 (Estimated); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Healthy; Obesity
MeSH Terms: conditions — Obesity | interventions — Ghrelin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ghrelin — 0.1 microgram/kg/min, intravenous for 60 minutes
  Other Names: Ghrelin (human) acetate

SUMMARY:
Ghrelin is a newly discovered peptide that is secreted by the stomach. Its main role is to stimulate food intake but recent studies indicate that it also acts on the cardiovascular system to confer beneficial effects. The mechanism of action is unclear but experimental studies suggest that ghrelin decreases the sympathetic nervous system. Beside there is new evidence in animal models that ghrelin may also be involved in stress reaction as ghrelin injection seems to protect against symptoms of stress. Given that circulating levels of ghrelin are reduced in obesity, this suggests that the effect of ghrelin may differ between lean and obese subjects. Ghrelin could represent an attractive therapeutic strategy for the treatment of cardiovascular diseases. The aim of the study if to gain more knowledge of the effect of ghrelin on the sympathetic nervous system and stress reactivity in both lean and obese subjects.

DETAILED DESCRIPTION:
This study will investigate the effect of intravenous administration of ghrelin on blood pressure, heart rate, muscle sympathetic nervous activity and baroreflex control in lean and obese individuals and will investigate whether ghrelin administration can influence the response to stress. Both lean and obese individuals will be recruited and will receive an intravenous administration of ghrelin at increasing doses for 1 hour. Their blood pressure, heart rate and sympathetic activity (small recording electrode in the peroneal nerve) will be recorded and subjects will be submitted to a mental arithmetic stress towards the end of the infusion. Blood samples will be taken at regular intervals for various metabolic tests. These responses will be compared to those when submitted to saline infusion.

ELIGIBILITY:
Inclusion Criteria:

* healthy lean subjects with a BMI < 25 kg/m2 and subjects with central obesity (according to IDF definition)

Exclusion Criteria:

* any current medication
* a history of diabetes
* hypertension
* cardiovascular, cerebrovascular, liver, thyroid disease
* mental illness

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2009-06; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Sympathetic nervous activity | 60 min

SECONDARY OUTCOMES:
blood pressure | 60 min

CONTACTS AND LOCATIONS:
Locations (1):
- Alfred & Baker Medical Unit, Melbourne, Victoria, Australia